CLINICAL TRIAL: NCT01400074
Title: A Phase III Multi-center, Open-label, Randomized Study of the Efficacy of Nilotinib Versus Imatinib in Adult Patients With Ph+ CML in Early CP Who Have a Suboptimal Molecular Response to Imatinib
Brief Title: Efficacy of Nilotinib Versus Imatinib in Ph+ CML in Early CP Who Have a Suboptimal Molecular Response to Imatinib
Acronym: RE-NICE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Dong-Wook Kim, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107AKR01T
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nilotinib (Active Comparator): 400 mg twice daily
  Interventions: Drug: Nilotinib, Imatinib
- Imatinib (Active Comparator): 400 mg twice daily
  Interventions: Drug: Nilotinib, Imatinib

INTERVENTIONS:
Drug: Nilotinib, Imatinib — Nilotinib: 400 mg twice daily Imatinib: 400 mg twice daily
  Other Names: Nilotinib (AMN107): Tasigna; Imatinib (STI571): Gleevec

SUMMARY:
In this study, the efficacy of nilotinib at 400 mg BID will be compared with imatinib at 400 mg BID in suboptimal molecular response patients. To determine study eligibility, suboptimal molecular response will be defined as patients who have achieved a complete cytogenetic response (CCyR) but have not achieved a MMR, after at least 18 months of treatment on first line imatinib therapy at a minimum dose of 400mg daily (Baccarani 2006).

DETAILED DESCRIPTION:
Imatinib mesylate (imatinib) binds to the inactive conformation of Bcr-Abl tyrosine kinase suppressing the Ph+ clone in CML (Giles et al, 2005). It is effective in CML and is a major advance in therapy. With standard dose imatinib, the MMR and complete molecular response (CMR) rates are 35% to 40% and 6% to 10% respectively at 12 months. These surrogate endpoints have been associated with high long term survival rates (Kantarjian et al, 2004).

For patients who had a CCyR and MMR (defined as a reduction in Bcr-Abl transcript levels of at least 3 log at 12 months following imatinib therapy), the probability of remaining progression-free was 100 percent at 24 months, compared with 95% for patients achieved a CCyR but no MMR and 85% for patients who did not achieve a CCyR (P<0.001) (Hughes et al, 2003/Druker et al, 2006).

With continued doses of imatinib 400 mg/day, MMR at 24 months is 54% (IRIS SmPC data), however with high dose imatinib 800 mg/day, MMR may be 70%. Higher doses of imatinib improved the CCyR rates to 90% both in patients who failed prior IFN-alfa therapy and in those previously untreated (Cortes et al, 2005). Higher doses are expected to yield higher MMR rates at 24 months (Cortes et al, ASH 2004 poster). There is also a continued increase in the cumulative major/complete cytogenetic and molecular response rates with therapy, even after 2 years (Kantarjian 2004).

Nilotinib is a novel, oral tyrosine kinase inhibitor with improved potency compared with imatinib. In pre-clinical models of imatinib-sensitive CML cell lines, nilotinib was 20-50 times more potent than imatinib, and 3-7 times more potent in imatinib-resistant cell lines. In a Phase I dose-escalation trial [Study CAMN107A2101], 119 imatinib-resistant Ph+ CML and ALL patients were treated with single oral doses of nilotinib ranging from 50-1200 mg daily or 400 mg and 600 mg given twice daily. Nilotinib produced high hematologic and cytogenetic response rates of 92% and 53%, respectively (CCyR in 35%), in patients with chronic phase CML, who were resistant to imatinib. Nilotinib was found to have an acceptable tolerability profile (Kantarjian et al, 2005). Preliminary results from an ongoing Phase II study appear to confirm the efficacy and safety profile of nilotinib (Kantarjian et al, 2006).

Achievement of a major molecular response is an important short-term goal in CML therapy as it appears to predict for long-term event-free survival. This study is designed to compare the efficacy of nilotinib 400 mg twice daily with patients' maximum tolerated doses of imatinib (optimally 800 mg/day) in producing a major molecular response after 12 months of treatment in individuals previously not in major molecular remission. It will also examine the rates of major molecular and complete molecular response in each of the treatment arms, as achievement of these endpoints may also be of prognostic significance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* ECOG 0, 1, or 2
* Diagnosis of Ph+ CML in CP
* Patients with suboptimal molecular response defined as:

  * Patients must achieve a CCyR at 12 months and must maintain CCyR until study entry (0% Ph+ chromosomes). Cytogenetic confirmation of Ph+ (9;22 translocation) is required on a minimum of 20 metaphases. FISH analysis will not be accepted.
  * at least 18 months and up to 24 months (≥18 to ≤24 months) of treatment with imatinib as first line therapy, at a dose of 400 mg daily, without achieving a MMR (<0.1% IS of Bcr-Abl transcript by RQ- PCR).
* The following laboratory results must be present:

  * Total bilirubin <1.5 x ULN
  * SGOT and SGPT <2.5 x ULN
  * Creatinine <1.5 x ULN
  * Serum amylase and lipase ≤ 1.5 x ULN
  * Alkaline phosphatase ≤ 2.5 x ULN unless considered tumor related.
  * Serum potassium, magnesium and calcium ≥ LLN or correctable with supplements to within normal limits prior to the first dose of study medication.
* Ability to provide written informed consent prior to any study related screening procedures being performed.

Exclusion Criteria:

* Late CP who started imatinib more than 6 months after diagnosis
* Prior accelerated phase or blast phase CML
* Rare hereditary problems of galactose intolerance, severe lactase deficiency or glucose galactose malabsorption
* Hypersensitivity to nilotinib or any of the excipients.
* Previously documented T315I mutations.
* Intolerance to imatinib 400 mg daily defined as the inability to maintain at least 400 mg daily for the previous 3 months.
* Patients treated with imatinib more than 400mg daily
* Achieved prior MMR or CCyR on imatinib and lost response to entering the study.
* Previous treatment with interferon or any other tyrosine kinase inhibitor except imatinib (however, allow hydroxyurea or anagrelide before initial imatinib start)
* Impaired cardiac function
* Treatment with inhibitors of CYP3A4 or medications well documented to prolong the QT interval are contraindicated
* Impaired gastrointestinal (GI) function or GI disease
* History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis.
* Known cytopathologically confirmed CNS infiltration (in absence of suspicion of CNS involvement, lumbar puncture not required).
* Any other malignancy that is clinically significant or requires active intervention.
* Severe or uncontrolled medical conditions (i.e. uncontrolled diabetes, acute or chronic liver disease, pancreatic, or severe renal disease unrelated to tumor, active or uncontrolled infection).
* History of significant congenital or acquired bleeding disorder unrelated to cancer.
* Previous radiotherapy to ≥ 25% of the bone marrow.
* Major surgery within 4 weeks prior to Day 1 of study or who have not recovered from prior surgery.
* Use of therapeutic coumarin derivatives (i.e. warfarin, acenocoumarol, phenprocoumon).
* Treatment with other investigational agents within 30 days of Day 1.
* History of non-compliance to medical regimens or inability to grant consent.
* Women who are pregnant, breast feeding, or of childbearing potential without a negative serum or urine pregnancy test at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
the cumulative rate of MMR | 12 months
  To evaluate the cumulative rate of MMR at 12 months of nilotinib compared to imatinib in adult patients with Ph+ CML in early CP who have suboptimal molecular response to imatinib

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Wook Kim, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea